CLINICAL TRIAL: NCT04995263
Title: A Multicomponent Intervention for Prevention and Treatment of Sleep Disturbances in a Psychiatric Intensive Care Unit: A Before-After, Randomized, Controlled Trial
Brief Title: A Multicomponent Intervention for Prevention and Treatment of Sleep Disturbances in a Psychiatric Intensive Care Unit
Acronym: SUEÑA-SM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: UC CHRISTUS (Unknown)
Responsible Party: Principal Investigator, Constanza Caneo, Clinical Assistant Professor, C-L Psychiatrist, SUEÑA Director, Pontificia Universidad Catolica de Chile
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 0
Record Dates: First submitted 2021-07-22; First posted 2021-08-06 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Dyssomnias
Keywords: Sleep; Psychiatric Intensive Care Unit; Multicomponent Intervention; Wearable Activity Tracker; Behavioral Intervention; Psychoeducation; Environmental Interventions
MeSH Terms: conditions — Dyssomnias | interventions — Ear Protective Devices

STUDY DESIGN:
Intervention Model Description: Before-after design for the implementation of unit-wide intervention, with a later randomization for individualized interventions.
Who Masked: Outcomes Assessor
Masking Description: Two investigators will work on-site collecting data for each of the variables, uploading them to a secure database (REDCap) as anonymous data. Afterwards, data and outcomes will be analyzed by a blinded investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pre-intervention, control group (No Intervention): A basal measurement of primary and secondary outcomes of the target population, prior to the implementation the intervention. Estimated duration 3 months, n = 30.
- Post-intervention, SUEÑA half bundle, active group 1 (Experimental): Post-intervention, environmental and behavioral modifications in patient care interventions.
  Implementation of components 1 through 4 of SUEÑA intervention in the entire PICU unit. All participants will be exposed to the intervention. Estimated duration: 3 months, n = 30.
  Interventions: Behavioral: Sueña component 1: Sleep Hygiene Promotion; Behavioral: Sueña component 2: Periodic Anxiety and Pain Screening; Behavioral: Sueña component 3: Hypnotics and Caffeine Regulation; Behavioral: Sueña component 4: Sleep Masks and Ear Plugs
- Post-intervention, randomization for SUEÑA half bundle plus, active group 2 (Experimental): Randomization for full SUEÑA bundle: environmental and behavioral modifications in patient care interventions plus sleep informed treatment.
  Participants will be randomized to receive SUEÑA components 1 through 5 Estimated duration: 6 months, n = 30
  Interventions: Behavioral: Sueña component 1: Sleep Hygiene Promotion; Behavioral: Sueña component 2: Periodic Anxiety and Pain Screening; Behavioral: Sueña component 3: Hypnotics and Caffeine Regulation; Behavioral: Sueña component 4: Sleep Masks and Ear Plugs; Other: Sueña component 5: Personalized Psychoeducation
- Post-intervention, randomization for SUEÑA full bundle, active group 3 (Experimental): Randomization for full SUEÑA bundle: environmental and behavioral modifications in patient care interventions plus sleep informed treatment and personalized psychoeducation.
  . Participants will be randomized to receive SUEÑA components 1 through 6. Estimated duration: 6 months, n = 30
  Interventions: Behavioral: Sueña component 1: Sleep Hygiene Promotion; Behavioral: Sueña component 2: Periodic Anxiety and Pain Screening; Behavioral: Sueña component 3: Hypnotics and Caffeine Regulation; Behavioral: Sueña component 4: Sleep Masks and Ear Plugs; Other: Sueña component 5: Personalized Psychoeducation; Device: Sueña component 6: Sleep Reports

INTERVENTIONS:
Behavioral: Sueña component 1: Sleep Hygiene Promotion — The nursery staff will be instructed to promote sleep hygiene. Nurse technicians will: inform patients of the efforts to ensure a healthy sleep environment, verify the minimization of light and noise after 23:00 PM, favour natural light after 07:00 AM, and foment patient's activities and participation in group therapy. Nurses will: reduce sleep interruptions to a minimum, to only perform actions (i.e. blood testing, clinical controls, medicine administration) deemed strictly necessary between 23:00 PM and 07:00 AM. A list of commonly used medications with their pharmacodynamic and pharmacokinetic properties tailored by a pharmaceutical chemist will be provided, to ensure optimal medication administration while protecting the guaranteed sleep hours, to be coordinated with the treating physician.
  Arms: Post-intervention, SUEÑA half bundle, active group 1; Post-intervention, randomization for SUEÑA full bundle, active group 3; Post-intervention, randomization for SUEÑA half bundle plus, active group 2
Behavioral: Sueña component 2: Periodic Anxiety and Pain Screening — Every night, nursery staff will include anxiety and pain screenings as part of vital signs assessments, using visual analog scales for each one. If any screening is altered, clinical actions will be performed to alleviate symptomatology if deemed necessary, using clinical judgement.
  Arms: Post-intervention, SUEÑA half bundle, active group 1; Post-intervention, randomization for SUEÑA full bundle, active group 3; Post-intervention, randomization for SUEÑA half bundle plus, active group 2
Behavioral: Sueña component 3: Hypnotics and Caffeine Regulation — The use of hypnotics will be standardized to be administered no later than at 22:00 PM; in the case of melatonin, its administration will be suggested at sundown, at 20:00 PM. Caffeinated drinks will be prohibited after 15:00 PM.
  Arms: Post-intervention, SUEÑA half bundle, active group 1; Post-intervention, randomization for SUEÑA full bundle, active group 3; Post-intervention, randomization for SUEÑA half bundle plus, active group 2
Behavioral: Sueña component 4: Sleep Masks and Ear Plugs — Sleep masks and ear plugs will be available to all patients if they wish to use them. The nursery team will reinforce its use between 23:00 PM and 07:00 AM.
  Arms: Post-intervention, SUEÑA half bundle, active group 1; Post-intervention, randomization for SUEÑA full bundle, active group 3; Post-intervention, randomization for SUEÑA half bundle plus, active group 2
Other: Sueña component 5: Personalized Psychoeducation — Two individualized, nurse-led psychoeducation PowerPoint presentations on sleep hygiene will be presented to patients, supported by educational material aimed at the patient and their families.
  Arms: Post-intervention, randomization for SUEÑA full bundle, active group 3; Post-intervention, randomization for SUEÑA half bundle plus, active group 2
Device: Sueña component 6: Sleep Reports — Objective and subjective reports of sleep quality will be handed to attending psychiatrist, using data gathered with wearable devices (Fitbit Charge 4) and self-report questionnaires regarding perceived sleepiness and overall sleep. The psychiatrist in charge uses said information in the routine case management
  Arms: Post-intervention, randomization for SUEÑA full bundle, active group 3

SUMMARY:
Hospitalized adult patients suffer from sleep deprivation, which has been associated with multiple negative consequences, both in short and in the long term. Many factors have been attributed to poor sleep quality, including excessive noise, inappropriate lighting, interactions with the healthcare team, administration of drugs, patients' symptoms, among others. There is scarce evidence reporting multicomponent interventions aimed at ensuring and improving sleep quality in hospitalized patients. The following before-after, randomized controlled trial will evaluate and determine the feasibility, acceptability and effectivity of a multicomponent intervention in improving sleep quality and reducing the consequences of poor sleep in a psychiatric intensive care unit (PICU). The intervention is comprised of changes in health personnel habits, improvements in the PICU environment, patient's psychoeducation and continuous sleep and activity monitoring through a validated wearable device.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in the last 72 hours.
* Capacity to consent
* Approval by treating physician

Exclusion Criteria:

* Active psychosis
* Active eating disorder
* Delirium
* Major cognitive disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-06-22 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Total Sleep Time | From enrollment, during the first 72 hours of hospitalization, for up to 14 days or discharge.
  Measured in hours and minutes, using objective data obtained via Fitbit Charge 4 devices, and subjective data obtained directly from the patient using the Sleep Diary, a consensus tool for the self report of different standardized sleep variables.

SECONDARY OUTCOMES:
Change in Mean Number and Total Duration of Nocturnal Awakenings | From enrollment, during the first 72 hours of hospitalization, for up to 14 days or discharge.
  Measured in integer numbers for mean number and minutes for duration, using subjective data obtained directly from the patient using the Sleep Diary, and objective data obtained via Fitbit Charge 4 devices.
Change in Mean Number and Total Duration of Naps During the Day | From enrollment, during the first 72 hours of hospitalization, for up to 14 days or discharge.
  Measured in integer numbers for mean number and minutes for duration, using subjective data obtained directly from the patient using the Sleep Diary, and objective data obtained via Fitbit Charge 4 devices.
Change in Average Time of Falling Sleep and Awakening | From enrollment, during the first 72 hours of hospitalization, for up to 14 days or discharge.
  Measured in time of day in 24-hour notation, using subjective data obtained directly from the patient using the Sleep Diary, and objective data obtained via Fitbit Charge 4 devices.
Change in Sleep Architecture | From enrollment, during the first 72 hours of hospitalization, for up to 14 days or discharge.
  Measured in minutes of total duration for each sleep phase (awake, light sleep, deep sleep and REM) and as a relative value of the total sleep time, using objective data measured by Fitbit Charge 4 devices.
Change in Sleep Onset Latency Mean Duration | From enrollment, during the first 72 hours of hospitalization, for up to 14 days or discharge.
  Measured in minutes of total time spent awake from the time of going to bed with the intention of falling asleep to the time of the first registered sleep phase, using subjective data from the Sleep Diary and objective data measured by Fitbit Charge 4 devices.
Change in REM Onset Latency Mean Duration | From enrollment, during the first 72 hours of hospitalization, for up to 14 days or discharge.
  Measured in minutes of total time spent awake from the time of going to bed with the intention of falling asleep to the time of the first registered REM phase, using subjective data from the Sleep Diary and objective data measured by Fitbit Charge 4 devices.
Change in Wake After Sleep Onset Mean Duration | From enrollment, during the first 72 hours of hospitalization, for up to 14 days or discharge.
  Measured in minutes of total time spent awake from the time of the first registered sleep phase to the time of the last registered awakening, using objective data measured by Fitbit Charge 4 devices.
Change in Sleep Efficiency | From enrollment, during the first 72 hours of hospitalization, for up to 14 days or discharge.
  Measured in percentage of total time spent sleeping at night, calculated as total sleep time divided by total time spent in bed, using subjective data from the Sleep Diary and objective data measured by Fitbit Charge 4 devices.
Change in Mean Heart Rate | From enrollment, during the first 72 hours of hospitalization, for up to 14 days or discharge.
  Measured in integer numbers, using objective data measured by Fitbit Charge 4 devices, considering the heart rate during the day and while in bed.
Change in Mean Number of Steps | From enrollment, during the first 72 hours of hospitalization, for up to 14 days or discharge.
  Measured in integer numbers, using objective data measured by Fitbit Charge 4 devices.
Change in Mean Level of Sound | From enrollment, during the first 72 hours of hospitalization, for up to 14 days or discharge.
  Measured in decibels, using objective data registered by a decibel meter placed in the participant's rooms.
Change in Mean Level of Light | From enrollment, during the first 72 hours of hospitalization, for up to 14 days or discharge.
  Measured in lux, using objective data registered by a lux meter placed in the participant's rooms.
Changes in Sleep Quality Perception | From enrollment, during the first 72 hours of hospitalization, for up to 14 days or discharge.
  Measured using the Richard Campbell Sleep Questionnaire (RCSQ), which considers 5 domains in Likert scales, and registers a mean score of all domains.
Changes in Daytime Sleepiness | From enrollment, during the first 72 hours of hospitalization, for up to 14 days or discharge.
  Measured using the Epworth Sleepiness Scale (ESS), which considers 8 hypothetical situations and scores the likelihood of falling asleep from 0 to 3, and registers a total aggregated score (with a maximum total score of 24).
Changes in Subjective Perception of Sleep-Disturbing Factors | From enrollment, during the first 72 hours of hospitalization, for up to 14 days or discharge.
  Measured using complementary questions regarding the presence/absence of factors (either environmental, symptomatological, or other) and their identification using predefined options: excessive light, excessive noise, interactions with health personnel, pain, anxiety, or others. In case of selecting "others", a text field will be available for its description.
Changes in Pharmacological Indications and Need of SOS Medication | From enrollment, during the first 72 hours of hospitalization, for up to 14 days or discharge.
  Registered using extensive charts of common use medications during hospitalization, obtaining data registered in the participant's daily medical chart.
Changes in Systolic and Diastolic Blood Pressure | From enrollment, during the first 72 hours of hospitalization, for up to 14 days or discharge.
  Measured in millimetres of mercury (mmHg), using morning data registered in the participant's daily medical chart.
Level of Pain | From enrollment, during the first 72 hours of hospitalization, for up to 14 days or discharge. To be measured from the second branch onward, after the environmental interventions implementation.
  Measured with a Visual Analog Scale for Pain (scores ranging from 0 - 10 points), using data registered at 20:00 PM, in the participant's daily medical chart.
Level of Anxiety | From enrollment, during the first 72 hours of hospitalization, for up to 14 days or discharge. To be measured from the second branch onward, after the environmental interventions implementation.
  Measured with a Visual Analog Scale for Anxiety (scores ranging from 0 - 10 points), using data registered at 20:00 PM, in the participant's daily medical chart.
Change in Mean Length of Stay | From day 1 of hospitalization until discharge
  Measured in days, using data from the participant's medical record.
Change in 30-day Readmission Rate | 30 days after the participant's discharge.
  Measured as a proportion, using data from the participant's medical record and telephonic follow-up.
Change in Participant Satisfaction Regarding Sleep During Hospitalization | 7 days after the participant's discharge.
  Measurement of the subjective experience of the participant, using telephone surveys.
Participant Satisfaction Regarding the Intervention | 7 days after the participant's discharge.
  Measurement of the subjective experience of participants, using telephone surveys.
Health Personnel Satisfaction and Agreeability Regarding the Intervention | Every 3 months through study completion, an average of 1.5 years
  Measurement of the subjective experience of treating physicians and nursery team, using web-based surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Constanza Caneo Robles, MD, Study Director — Pontifica Universidad Católica de Chile; Juan C Rodríguez, MD, Study Director — Pontifica Universidad Católica de Chile; María Rodríguez Fernández, PhD, Study Chair — Pontifica Universidad Católica de Chile; Marcela Babul, MD, Study Chair — Pontifica Universidad Católica de Chile
Locations (1):
- Clínica San Carlos de Apoquindo UC, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Yes
We are available to be contacted by researchers aiming to conduct secondary analyses based on our study, after providing a study protocol based on international guidelines, in order to ensure adequate use of our data.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: January 2024
Access Criteria: contact to responsable researcher C Caneo

REFERENCES:
- [Background] Bano M, Chiaromanni F, Corrias M, Turco M, De Rui M, Amodio P, Merkel C, Gatta A, Mazzotta G, Costa R, Montagnese S. The influence of environmental factors on sleep quality in hospitalized medical patients. Front Neurol. 2014 Dec 11;5:267. doi: 10.3389/fneur.2014.00267. eCollection 2014. PMID 25566173
- [Background] Bernhofer EI, Higgins PA, Daly BJ, Burant CJ, Hornick TR. Hospital lighting and its association with sleep, mood and pain in medical inpatients. J Adv Nurs. 2014 May;70(5):1164-73. doi: 10.1111/jan.12282. Epub 2013 Oct 27. PMID 24164506
- [Background] Bourne RS, Mills GH. Sleep disruption in critically ill patients--pharmacological considerations. Anaesthesia. 2004 Apr;59(4):374-84. doi: 10.1111/j.1365-2044.2004.03664.x. PMID 15023109
- [Background] Denkinger MD, Lindemann U, Nicolai S, Igl W, Jamour M, Nikolaus T. Assessing Physical Activity in Inpatient Rehabilitation: validity, practicality, and sensitivity to change in the physical activity in inpatient rehabilitation assessment. Arch Phys Med Rehabil. 2011 Dec;92(12):2012-7. doi: 10.1016/j.apmr.2011.06.032. PMID 22133250
- [Background] Horne S, Hay K, Watson S, Anderson KN. An evaluation of sleep disturbance on in-patient psychiatric units in the UK. BJPsych Bull. 2018 Oct;42(5):193-197. doi: 10.1192/bjb.2018.42. PMID 30229719
- [Background] Hu RF, Jiang XY, Chen J, Zeng Z, Chen XY, Li Y, Huining X, Evans DJ. Non-pharmacological interventions for sleep promotion in the intensive care unit. Cochrane Database Syst Rev. 2015 Oct 6;2015(10):CD008808. doi: 10.1002/14651858.CD008808.pub2. PMID 26439374
- [Background] Kanji S, Mera A, Hutton B, Burry L, Rosenberg E, MacDonald E, Luks V. Pharmacological interventions to improve sleep in hospitalised adults: a systematic review. BMJ Open. 2016 Jul 29;6(7):e012108. doi: 10.1136/bmjopen-2016-012108. PMID 27473952
- [Background] Lawrence G, Muza R. Assessing the sleeping habits of patients in a sleep disorder centre: a review of sleep diary accuracy. J Thorac Dis. 2018 Jan;10(Suppl 1):S177-S183. doi: 10.21037/jtd.2017.12.127. PMID 29445542
- [Background] Milani RV, Bober RM, Lavie CJ, Wilt JK, Milani AR, White CJ. Reducing Hospital Toxicity: Impact on Patient Outcomes. Am J Med. 2018 Aug;131(8):961-966. doi: 10.1016/j.amjmed.2018.04.013. Epub 2018 May 3. PMID 29729240
- [Background] Pilkington S. Causes and consequences of sleep deprivation in hospitalised patients. Nurs Stand. 2013 Aug 7-13;27(49):35-42. doi: 10.7748/ns2013.08.27.49.35.e7649. PMID 23924135
- [Background] Rodriguez JC, Dzierzewski JM, Alessi CA. Sleep problems in the elderly. Med Clin North Am. 2015 Mar;99(2):431-9. doi: 10.1016/j.mcna.2014.11.013. Epub 2014 Dec 30. PMID 25700593
- [Background] Sandoval-Rincon M, Alcala-Lozano R, Herrera-Jimenez I, Jimenez-Genchi A. [Validation of the Epworth sleepiness scale in Mexican population]. Gac Med Mex. 2013 Jul-Aug;149(4):409-16. Spanish. PMID 23999632
- [Background] Stewart NH, Arora VM. Sleep in Hospitalized Older Adults. Sleep Med Clin. 2018 Mar;13(1):127-135. doi: 10.1016/j.jsmc.2017.09.012. Epub 2017 Nov 10. PMID 29412979
- [Background] Tamrat R, Huynh-Le MP, Goyal M. Non-pharmacologic interventions to improve the sleep of hospitalized patients: a systematic review. J Gen Intern Med. 2014 May;29(5):788-95. doi: 10.1007/s11606-013-2640-9. Epub 2013 Oct 10. PMID 24113807
- [Background] Tembo AC, Parker V. Factors that impact on sleep in intensive care patients. Intensive Crit Care Nurs. 2009 Dec;25(6):314-22. doi: 10.1016/j.iccn.2009.07.002. Epub 2009 Oct 31. PMID 19880319
- [Background] Tullmann DF, Dracup K. Creating a healing environment for elders. AACN Clin Issues. 2000 Feb;11(1):34-50; quiz 153-4. doi: 10.1097/00044067-200002000-00006. PMID 11040551
- [Background] Wesselius HM, van den Ende ES, Alsma J, Ter Maaten JC, Schuit SCE, Stassen PM, de Vries OJ, Kaasjager KHAH, Haak HR, van Doormaal FF, Hoogerwerf JJ, Terwee CB, van de Ven PM, Bosch FH, van Someren EJW, Nanayakkara PWB; "Onderzoeks Consortium Acute Geneeskunde" Acute Medicine Research Consortium. Quality and Quantity of Sleep and Factors Associated With Sleep Disturbance in Hospitalized Patients. JAMA Intern Med. 2018 Sep 1;178(9):1201-1208. doi: 10.1001/jamainternmed.2018.2669. PMID 30014139
- [Result] Novak C, Packer E, Paterson A, Roshi A, Locke R, Keown P, Watson S, Anderson KN. Feasibility and utility of enhanced sleep management on in-patient psychiatry wards. BJPsych Bull. 2020 Dec;44(6):255-260. doi: 10.1192/bjb.2020.30. PMID 32329430